CLINICAL TRIAL: NCT05343845
Title: Does Smoking Effect Spinal Anesthesia in Parturient Women? A Randomized-controlled Trial
Brief Title: Does Smoking Effect Spinal Anesthesia?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hacı Yusuf Güneş, Assistant proffesor, Yuzuncu Yil University
Other Study IDs: 2019/18
Record Dates: First submitted 2022-02-28; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Smoking Cigarette; Spinal Anaesthesia; Pregnancy; Cesarean Section
Keywords: Spinal anesthesia; Cesarean section; Pregnant women; Smoking
MeSH Terms: conditions — Cigarette Smoking; Smoking | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group NS, Nonsmoker (n= 50): Pregnant women who did not smoke during pregnancy will be separated as Group NS. Local anesthetic dose adjusted for height and weight and 20 µg fentanyl will be administered intrathecally. Results regarding the effectiveness of spinal anesthesia will be monitored.
  Interventions: Other: Observational study
- Group S, Smoker (n= 50): Pregnant women who smoked 5 or more cigarettes in a day will be separated as Group S. A local anesthetic dose adjusted for height and weight and 20 µg fentanyl will be administered intrathecally. Results regarding the effectiveness of spinal anesthesia will be monitored.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — After approval of the institution's ethics committee, 100 patients will be divided in two groups as pregnant women who did not smoke during pregnancy and pregnant women who smoked 5 or more cigarettes in a day. The local anesthetic, which dose will adjusted according to height and weight, and 20 µg fentanyl will be administered intrathecally to both groups. Results on the effectiveness of spinal anesthesia will be monitored.

SUMMARY:
Background In the last 10 years, the rate of smoking in women of childbearing age has increased gradually. The smoking affects general anesthesia negatively. Can smoking also affect regional anesthesia in pregnant women? Our aim in this study is to investigate the effects of smoking on spinal anesthesia applied for C/S in pregnant women.

Methods After approval of the institution's ethics committee, 100 patients will divided in two groups as pregnant women who did not smoke during pregnancy and pregnant women who smoked 5 or more cigarettes in a day. The local anesthetic, which dose will be adjusted according to height and weight, and 20 µg fentanyl will administered intrathecally to both groups. Results on the effectiveness of spinal anesthesia will monitored.

Results The data of 100 parturients will investigated. The onset time of sensory and motor block, the duration of motor and sensory block, APGAR and VAS scores will be monitored. In addition, C/S indications, side effects, patient satisfaction, additional medication need and, spinal anesthesia preferences will be monitored.

Conclusions Smoking affects many systems. According to the onset of sensory block, duration of sensory and motor block and, VAS scores, which determine the effectiveness of spinal anesthesia, it will be evaluated whether smoking also affects spinal anesthesia in pregnant women.

DETAILED DESCRIPTION:
MATERIALS AND METHODS

Ethical approval:

This prospective, randomized-controlled, observational study was conducted at Van Research and Training Hospital with a bed capacity of 1500 located in Van, Turkey. Approval was obtained from the institution's ethics committee (2019/18), and the study was performed according to the World Medical Association's Declaration of Helsinki. All enrolled patients provided written informed consent.

Groups and Randomization: The patients included in the study will be divided into two groups. Pregnant women who did not smoke during pregnancy (Group NS, Non-Smoker) (n=50) and pregnant women who smoked 5 or more cigarettes per day (Group S, Smoker) (n=50) will be randomly included in the study.

Procedure: 8-10 mL/kg of crystalloid fluid intravenous hydration will be administered for 10-15 minutes to each patient taken to the operating table. Electrocardiography (ECG), peripheral oxygen saturation (SpO2) and noninvasive blood pressure (NIBP) monitoring will be routinely performed. NIBP values, heart rate (HR), and SpO2 values will be recorded before the procedure (T0).

After proper skin cleansing and sterile preparation with povidone-iodine, spinal anesthesia will be performed in a sitting position with a 25 gauge Quincke spinal needle at L3-4/4-5 level. After free cerebrospinal fluid (CSF) flow is seen, 7.5-10 mg heavy 0.5% (Marcaine spinal heavy, AstraZeneca PLC, Istanbul, Turkey) and 20 µg fentanyl (fentanyl 0.05 mg/ml, Johnson and Johnson, Istanbul, Turkey) ) will be administered intrathecally. Local anesthetic dose will be adjusted according to height and weight. Until the beginning of the surgical procedure, patients will be placed in a supine position with their heads slightly elevated and the operating table facing 15-20 degrees to the left to minimize aortocaval compression. The sensory block levels of the patients will be evaluated with the cold-hot test, and the motor block levels will be evaluated with the Bromage Scale at 2-minute intervals for the first 10 minutes. After intrathecal drug administration, the 1st (T1), 2nd (T2), 3rd (T3), 4th (T4), 5th (T5), 10th (T6), 15th (T7), 20th, and thirtieth Within minutes, hemodynamic parameters and SpO2 values will be recorded.

The onset time of sensory block: Time taken for the sensory block to reach the T6 dermatome.

The onset time of motor block: Time taken for the motor block to reach a Bromage score of 3.

After the adequate level of sensory block was achieved (thoracic 4-6 dermatome levels), the surgical procedure would be started. All patients will be given oxygen at a rate of 3 L/min with a face mask.

Duration of motor block: The overall duration of motor block was defined as the start of the motor block to the time when the motor block regressed to the level of 0 according to the Bromage Scale.

Duration of sensory block: The overall duration of sensory block was defined as the start of the sensory block to the time when the sensory block regressed to the level of the L1 dermatome. Sensory and motor block levels will be checked every 15 minutes intraoperatively and postoperatively, and sensory and motor block times will be recorded.

The time between the surgical incision and the clamping of the umbilical cord will be recorded. After the delivery of the newborn and the removal of the placenta, 20 IU of synthetic oxytocin will be infused in 1000 mL of crystalloid fluid. If needed, one ampoule of methylergonovine will administered intramuscularly (im). The patients who had discomfort during peritoneal irritation will sedated with fentanyl (50 mcg) and/or propofol, and the medications that were used will be recorded. Metoclopramide (10 mg) and ranitidine (50 mg) will administered intravenous to the patients with complaints of nausea and vomiting.

A decrease in MAP by more than 20% from the baseline or a decrease in MAP below 65 mmHg in the intraoperative period will considered as hypotension, and iv bolus of ephedrine (10 mg) will administered. The amount of ephedrine used during the operation will be recorded. When the heart rate fell below 50 beats/min, it will considered as bradycardia, and 0.5-0.75 mg of iv atropine will administered. A decrease in SpO2 below 90% will considered as low peripheral oxygen saturation, and the amount of oxygen given to these patients by a facemask will increased to 4-5 L/min.

Side effects such as nausea, vomiting, headache, chest pain, hypotension, and bradycardia will be recorded. The 1st- and 5th-minute APGAR scores of the newborns will be recorded. The satisfaction level of the patients (scored as not satisfied, less satisfied, very satisfied) will be recorded. The time between the beginning of the surgical incision and the last suture to close the skin will be recorded as the operation duration. The patients will be informed about the Visual Analogue Scale, which would be used to evaluate the pain they felt preoperatively, intraoperatively and postoperatively (0: No pain - 10: extreme pain). In the postoperative period, if the VAS score will 4 or higher, 1000 mg paracetamol will be administered intravenously for analgesia.

Statistical analysis: The statistical analyses will be performed using the Statistical Package for the Social Sciences 27.0 software for Windows (SPSS, Chicago, IL, USA).

Descriptive statistics will be presented as mean, standard deviation, median, minimum, maximum, frequency and percentage values. The distributions of the variables will evaluated with Kolmogorov-Smirnov test. Independent-samples t-test and Mann-Whitney U test will be used in the analyses of the quantitative data in independent groups. Chi-squared test will be used in the analyses of the qualitative data in independent groups, and Fisher's test will be used when the chi-squared test conditions were not met.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an American Society of Anesthesiologists (ASA) status of class I-II,
* Aged between 18 and 45 years,
* Scheduled to undergo spinal anesthesia for elective C/S

Exclusion Criteria:

* The requirement of emergency C/S for delivery,
* ASA class ≥ III patients,
* A contraindication for spinal anesthesia,
* Multiple gestations,
* Placental abnormalities
* Allergy to local anesthetics,
* Height shorter than 150 cm,
* Coagulation disorders and
* Refusal of spinal anesthesia.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Aged between 18 and 45 years, scheduled to undergo spinal anesthesia for elective C/S will be included in this study. Pregnancy is a woman-specific condition.
Study Population: The data of 100 parturients will be investigated.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Sensory block onset, | The sensory block onset will assessed 3 min after administering the spinal anesthetic, up to 10 minute.
  After intrathecal drug administration, sensory block levels will be checked with cold-hot test per one-minute intervals in the first 10 minutes. Time taken for sensory block to reach T6 dermatome will be recorded.
Duration of motor block, | The motor block will be followed until Bromage scales regress to zero point, up to 6 hour.
  Motor block levels will be checked with the Bromage Scale every minute for the first 10 minutes after intrathecal drug administration.
  Overall duration of motor block was defined as the start of the motor block to the time when the motor block regresses to 0 level according to the Bromage scale.The motor block test will be repeated every 15 minutes during and after surgery until the Bromage Scale regresses to 0 point.
Duration of sensory block, | The duration of sensory block will be controlled until it regresses to the L1 level, up to 6 hour.
  After intrathecal drug administration, sensory block levels will be checked with cold-hot tes at 2-minute intervals in the first 10 minutes. The cold-hot test will be repeated every 15 minutes during and after surgery until the the sensory block regressed to the level of the L1 dermatome. Overall duration of sensory block was defined as the start of the sensory block to the time when the sensory block regresses to L-1 dermatome level.
VAS scores | Pain level will be checked with VAS score at 4-hour intervals up to 24 hours.
  Patients will be informed about the Visual Analogue Scale, which will be used to evaluate the pain they felt preoperatively, intraoperatively and postoperatively (0; No pain - 10; extreme pain).

CONTACTS AND LOCATIONS:
Overall Officials: Hacı Yusuf YG Güneş, Assist.prof, Principal Investigator — Van Yüzüncü Yıl University, Van Research and Training Hospital, Van, Turkey
Locations (1):
- Van Yüzüncü Yıl University, Faculty of Medicine, Van, Tusba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be share for other researchers
Supporting Information: Study Protocol, SAP
Time Frame: One year
Access Criteria: The access can be provided via the e-mail addresses below. hyusufgunes@hotmail.com nyuzkat@gmail.com

REFERENCES:
- [Background] Oncken C, Dornelas EA, Kuo CL, Sankey HZ, Kranzler HR, Mead EL, Thurlow MSD. Randomized Trial of Nicotine Inhaler for Pregnant Smokers. Am J Obstet Gynecol MFM. 2019 Mar;1(1):10-18. doi: 10.1016/j.ajogmf.2019.03.006. Epub 2019 Mar 27. PMID 31380506
- [Background] Dias-Dame JL, Cesar JA. Disparities in prevalence of smoking and smoking cessation during pregnancy: a population-based study. Biomed Res Int. 2015;2015:345430. doi: 10.1155/2015/345430. Epub 2015 May 14. PMID 26075231
- [Background] Al-Noori NM, Ibraheem NS, Abdulmunem MM. The impact of cigarette smoking on the efficiency of local anesthesia during simple tooth extraction. Saudi Dent J. 2021 Nov;33(7):674-678. doi: 10.1016/j.sdentj.2020.04.011. Epub 2020 May 7. PMID 34803318